CLINICAL TRIAL: NCT03963336
Title: D-dimer and the Use of Anticoagulation in IIH
Brief Title: Quantitative D-dimer Level and Anticoagulant Therapy in Idiopathic Intracranial Hypertension
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Sherine El Mously, Assistant Professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M201
Record Dates: First submitted 2019-05-15; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: IIH; D-dimer; microthrombi; anticoagulation
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Heparin, Low-Molecular-Weight; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): 12 IIH patients for whom serum D-dimer was assessed by ELISA.They received acetazolamide and anticoagulant LMWH in the prophylactic dose for 2 weeks then continued on acetazolamide. Follow up after 1 and 6 months through HIT6 test and ophthalmological assessment (visual acuity, Frisen classification for papilledema, visual field, and visual evoked potentials)
  Interventions: Drug: LMWH; Drug: acetazolamide
- Group B (Active Comparator): 12 IIH patients for whom serum D-dimer was assessed by ELISA. They received acetazolamide only. Follow up after 1 and 6 months through HIT6 test and ophthalmological assessment (visual acuity, Frisen classification for papilledema, visual field, and visual evoked potentials)
  Interventions: Drug: acetazolamide
- Control group (No Intervention): 24 healthy subjects for whom serum D-dimer was assessed by ELISA.

INTERVENTIONS:
Drug: LMWH — Subcutaneous LMWH 1mg/kg/day for 2 weeks
  Other Names: Clexan
  Arms: Group A
Drug: acetazolamide — Carbonic anhydrase inhibitor 1-2g/day for 6 months
  Other Names: Diamox
  Arms: Group A; Group B

SUMMARY:
Idiopathic intracranial hypertension (IIH) is a syndrome characterized by elevated intracranial pressure (ICP) of unknown etiology.

The investigators aim to study the quantitative D-dimer level and the role of anticoagulant therapy in the absence of occlusive sinus thrombosis in IIH patients.

DETAILED DESCRIPTION:
24 patients with IIH according to the modified Dandy criteria were enrolled. Headache impact test (HIT6), ophthalmological assessment including Frisen classification for papilledema, visual acuity, visual field by perimetry, and visual evoked potentials were performed to the patients.

Serum quantitative D-dimer level was measured using the enzyme-linked immunosorbent assay (ELISA) technique for the patients and for 24 healthy matched controls.

Patients were divided into two groups: group (A) received acetazolamide and low molecular weight heparin (LMWH) in a prophylactic dose for 2 weeks while group (B) received acetazolamide only. Both groups continued the acetazolamide 1-2g/day for 6 months.

The investigators followed-up the patients after one and six months later through the HIT6 test and the ophthalmological assessment.

ELIGIBILITY:
Inclusion Criteria:

* IIH patients of both sexes fulfilling the modified Dandy criteria

Exclusion Criteria:

* disturbed conscious level, focal neurological signs, seizures, cerebral venous sinus thrombosis or stenosis, deep venous thrombosis or pulmonary embolism, malignancy, and acute nephritic syndrome.
* Patients with signs of disseminated intravascular coagulopathy and septic sinus thrombosis
* patients with a history of cerebral granuloma or infection, cerebrovascular stroke, head trauma or surgery.
* pregnant females or those who terminated their pregnancy in the last four weeks were also excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
serum quantitative D-dimer | Baseline assessment
  higher serum D-dimer levels will be detected in IIH patients of both groups compared to controls

SECONDARY OUTCOMES:
HIT6 score | 1 and 6 months
  The HIT6 score will improve in both groups (A and B) after receiving the treatment (either acetazolamide or LMWH)
Frisen classification for papilledema | 6 months
  papilledema will improve in both groups (A and B) after receiving the treatment (either acetazolamide or LMWH)
Visual acuity (Log Mar) | 6 months
  Visual acuity will improve in both groups (A and B) after receiving the treatment (either acetazolamide or LMWH)
Visual field (Perimetry) | 6 months
  Visual field will improve in both groups (A and B) after receiving the treatment (either acetazolamide or LMWH)
Visual Evoked Potentials (VEP) | 6 months
  VEP will improve in both groups (A and B) after receiving the treatment (either acetazolamide or LMWH)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No